CLINICAL TRIAL: NCT03814941
Title: To Evaluate the Incidence of Artifacts in the Locally Developed AIMS Database.
Brief Title: The Incidence of Artifacts in the Anesthesia Information Management System Database.
Status: Completed | Type: Observational
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Chien-Chung,Huang, Official Title: Principal Investigator,Attending physician of anesthesiology, Mackay Memorial Hospital
Other Study IDs: 19MMHIS017e
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Artifacts; Integrated Advanced Information Management Systems
Keywords: Artifacts; anesthesia information management system

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- paper-based anesthesia record: The AIMS sampled the vital signs from the monitor every minute and stored in the database.
  The incidence of artifacts in the AIMS database was evaluated by paper-based documented anesthesia record.
  Interventions: Other: paper-based anesthesia record
- electronic documents: The AIMS sampled the vital signs from the monitor every minute and stored in the database.
  The incidence of artifacts in the AIMS database was evaluated by electric documented anesthesia record.
  Interventions: Other: electronic documents

INTERVENTIONS:
Other: paper-based anesthesia record — to evaluate the incidence of artifacts in the AIMS database by paper-based anesthesia record
  Groups: paper-based anesthesia record
Other: electronic documents — to evaluate the incidence of artifacts in the AIMS database by electronic documents anesthesia record
  Groups: electronic documents

SUMMARY:
The purpose of the study is to evaluate the incidence of artifacts in the developed AIMS database

DETAILED DESCRIPTION:
At first, the authors evaluated the accuracy of the traditional, manually completed paper-based documentation, which sets a benchmark for the accuracy that the electronic documentation and database provides.

At the second portion, the investigators used the paper-based documentation as a standard to compare the electronic documentation. The incidence of artifact was double checked by two investigators.

At the third portion, the authors calculated the artifact incidence in the AIMS database, using paper based and electric document anesthesia records as the standard respectively.

ELIGIBILITY:
Inclusion Criteria:

* patient undergo general or regional anesthesia
* elective surgery

Exclusion Criteria:

* emergency operation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients undergo general or regional anesthesia for surgery
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
percentage of artifacts | intraoperative (from the beginning to the end of anesthesia record)
  to evaluate how many percentage of artifacts for each of the included parameters

SECONDARY OUTCOMES:
deviating values | intraoperative (from the beginning to the end of anesthesia record)
  to calculate the number of values deviating from the predefined baseline value
percentage of devotional artifacts | intraoperative (from the beginning to the end of anesthesia record)
  to evaluate how many percentage of the deviations are artifacts
episodes of artifacts | intraoperative (from the beginning to the end of anesthesia record)
  to find out the average of number of episodes across each artifact
causes of artifacts | intraoperative (from the beginning to the end of anesthesia record)
  to find out the cause of the artifact and respective percentage

CONTACTS AND LOCATIONS:
Overall Officials: Chien-Chung Huang, MD, Study Director — Mackay Memorial Hospital
Locations (1):
- MacKay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilbanks BA, Berner ES, Alexander GL, Azuero A, Patrician PA, Moss JA. The effect of data-entry template design and anesthesia provider workload on documentation accuracy, documentation efficiency, and user-satisfaction. Int J Med Inform. 2018 Oct;118:29-35. doi: 10.1016/j.ijmedinf.2018.07.006. Epub 2018 Jul 24. PMID 30153918
- [Background] Kool NP, van Waes JA, Bijker JB, Peelen LM, van Wolfswinkel L, de Graaff JC, van Klei WA. Artifacts in research data obtained from an anesthesia information and management system. Can J Anaesth. 2012 Sep;59(9):833-41. doi: 10.1007/s12630-012-9754-0. Epub 2012 Jul 18. PMID 22806063
- [Background] Hoorweg AJ, Pasma W, van Wolfswinkel L, de Graaff JC. Incidence of Artifacts and Deviating Values in Research Data Obtained from an Anesthesia Information Management System in Children. Anesthesiology. 2018 Feb;128(2):293-304. doi: 10.1097/ALN.0000000000001895. PMID 28968279